CLINICAL TRIAL: NCT04139577
Title: Fecal Microbiota Transplantation (FMT) in for the Treatment of High-Risk Acute Graft-Versus-Host Disease (GVHD) After Allogeneic Hematopoietic Cell Transplantation (HCT)
Brief Title: FMT In High-Risk Acute GVHD After ALLO HCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Zachariah Michael DeFilipp, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-359
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Acute Graft-Versus-Host Disease (Gvhd) Grade; Hematopoietic Cell Transplantation; Fecal Microbiota Transplant
Keywords: Acute Graft-Versus-Host Disease (Gvhd) Grade; Hematopoietic Cell Transplantation; Fecal Microbiota Transplant
MeSH Terms: conditions — Graft vs Host Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fecal Microbiota Transplant (FMT) FOR HIGH-RISK ACUTE GVHD (Experimental): The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.
  this research study for up to 6 months. You may receive up to 2 cycles of the study treatment.
  - Fecal Microbiota Transplant ( FMT)- Oral Study Drug, predetermined dosage and timings, up to 2 cycles.
  * One cycle of treatment consists of one induction week of FMT followed by three weeks of maintenance FMT.
  * The maintenance weeks happen for 3 weeks after the induction week.
  * All doses will be administered in the clinic.
  * A second cycle of treatment as deemed appropriate
  Interventions: Biological: Fecal Microbiota Transplant

INTERVENTIONS:
Biological: Fecal Microbiota Transplant — FMT- Oral Study Drug, predetermined dosage and timings, up to 2 cycles
  Other Names: FMT

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Fecal Microbiota Transplant (FMT) treatment in high-risk acute graft-versus-host disease (GVHD).

This research study involves an experimental intervention called FMT.

DETAILED DESCRIPTION:
In this research study, the investigators are evaluating the effectiveness of Fecal Microbiota Transplant (FMT) treatment in high-risk acute GVHD. The investigators are evaluating the effectiveness of FMT (also known as 'stool transplantation' or 'fecal transplant') in being able to transfer gut organisms from a healthy donor to the patient.

The investigators are also evaluating the ability of this treatment to improve or completely resolve the clinical symptoms (diarrhea, abdominal pain, rash, liver inflammation) that can occur with acute GVHD.This research study is a Pilot Study, which is the first time investigators are examining this intervention for treatment of acute GVHD.

The FDA (the U.S. Food and Drug Administration) has not approved FMT for this use. The FDA has classified human stool as a biological agent and determined that its use in FMT therapy should be regulated to ensure patient safety. To use FMT to treat recurrent Clostridium difficile infection, the most common indication for FMT, does not require an investigation new drug permit. To use FMT for research or to treat any condition other than recurrent Clostridium difficile infection requires an investigation new drug permit. An investigation new drug permit has been obtained for this study.

* After HCT, the body's microbiome (the natural existence of various bacteria and organisms) in the intestinal tract may be affected, in that the number and types of good bacteria is reduced (also called a reduction in microbial flora diversity). Studies have shown that the number and types of good bacteria in the gut can impact whether or not graft-versus-host disease (GVHD) is developed. GVHD occurs when donated bone marrow cells attack the body with an immune response.
* FMT is a process utilizing microbial components which are the good, healthy bacteria that would otherwise naturally occur the body. Since may have decreased microbial flora diversity after HCT, these microbial components are taken from a stool donor. They are extracted from fecal matter (stool) and put into a capsule to ingest.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years old
* Patient has undergone allogeneic hematopoietic cell transplantation from any donor (related or unrelated with any degree of HLA matching) and any donor source (bone marrow, peripheral blood stem cells, or cord blood) for a hematologic malignancy or disorder. Recipients of myeloablative and reduced-intensity conditioning regimens are eligible.
* Evidence of myeloid engraftment (eg, absolute neutrophil count ≥ 0.5 × 109/L for 3 consecutive assessments if ablative therapy was previously used). Use of growth factor supplementation is allowed.
* Patient must have clinically suspected Grade II to IV aGVHD as per MAGIC criteria. Clinical suspicion of aGVHD by the treating physician is sufficient and biopsies are not required to pathologically confirm aGVHD. However, in situations where alternative diagnoses of drug effects or infection are not adequately ruled out on clinical suspicion alone, biopsies are recommended. - Patients must have a diagnosis of high-risk acute GVHD, defined as either:

  -- Steroid-refractory GVHD:
  * Progressive GVHD after at least 3 days of systemic corticosteroids (≥ 1 mg/kg/day of prednisone equivalent), OR
  * No improvement in GVHD after at least 7 days on ≥ 1 mg/kg/day of prednisone equivalent or insufficient improvement which warrants the addition of another agent, OR
  * Flare of GVHD symptoms during taper.
* High-risk, treatment-naïve GVHD

  * AA3 risk by Ann Arbor GVHD scoring risk system
  * Treatment-naïve: less than 3 days of therapy with systemic corticosteroids (≥ 1 mg/kg/day of prednisone equivalent)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for 3 months after FMT.
* Ability to understand and the willingness to sign a written informed consent document, including the willingness to accept risk of unrelated donor stool.
* Ability to swallow large capsules.

Exclusion Criteria:

* Participants who have initiated a new systemic treatment for steroid-refractory GVHD (institutional standard or investigational agent) within the 2 weeks prior to first dose of FMT. Treatment with FMT is allowed once the time since initiation of newest systemic therapy is 2 weeks or longer.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Delayed gastric emptying syndrome or large hiatal hernia
* Known chronic aspiration
* Participants with a history of significant allergy to foods not excluded from the donor diet (excluded foods are tree nuts, peanuts, shellfish, eggs)
* Pregnant and breast-feeding women are ineligible because they are not eligible for hematopoietic stem cell transplantation.
* HIV-positive participants are ineligible.
* Participants who are unable to swallow pills.
* Participants with end-stage liver disease (cirrhosis)
* Participants with acute, active gastrointestinal infection (e.g., typhlitis, diverticulitis, appendicitis)
* Participants with inflammatory bowel disease (e.g., ulcerative colitis, Crohn's)
* Prior total colectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are able to swallow ≥ 40 capsules (out of 75) | 29 Days
  Based on this information, FMT will be considered feasible if, among the 11 eligible patients, ≥8 patients are able to swallow ≥ 40 capsules.

SECONDARY OUTCOMES:
Response Rate-Acute GVHD | 29 Days
  Kaplan-Meier estimates
Overall Survival | 6 months, 12 Months
  Kaplan-Meier estimates
Progression Free Survival | 6 months, 12 Months
  Kaplan-Meier estimates
Non-relapse mortality (NRM) | 6 month, 12 Months
  time from first dose of FMT to death without relapse or progression or underlying disease. Deaths from any cause without prior progression are considered as NRM events

CONTACTS AND LOCATIONS:
Overall Officials: Zachariah DeFilipp, MD, Principal Investigator — Masachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to the Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] DeFilipp Z, Damania AV, Kim HT, Chang CC, El-Jawahri A, McAfee SL, Bottoms AS, Toncheva V, Smith MM, Dolaher M, Perry L, White M, Diana B, Connolly S, Dey BR, Frigault MJ, Newcomb RA, O'Donnell PV, Spitzer TR, Mansour MK, Weber D, Ajami NJ, Hohmann E, Jenq RR, Chen YB. Third-party fecal microbiota transplantation for high-risk treatment-naive acute GVHD of the lower GI tract. Blood Adv. 2024 May 14;8(9):2074-2084. doi: 10.1182/bloodadvances.2024012556. PMID 38471063